CLINICAL TRIAL: NCT06507163
Title: The Effect of Breathing Exercise Applied With Incentive Spirometer on Pain, Anxiety, Comfort and Physiological Parameters Before and After Surgery in Cardiac Surgery Patients
Brief Title: The Effect of Breathing Exercise Applied With Incentive Spirometer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut, Associate Prof., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2318
Record Dates: First submitted 2024-07-06; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Breathing Exercises; Cardiac Surgery; Incentive Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The post-surgical breathing exercise group (Experimental): Individuals in this group were asked to perform 10 breathing exercises with IS every waking hour in addition to the routine practices of the clinic for 5 days in the postoperative period.
  Interventions: Other: The post-surgical breathing exercise group
- The pre- and post- surgical breathing exercise group (Experimental): Individuals in this group were asked to perform 10 breathing exercises with IS every waking hour in addition to the routine practices of the clinic for a total of 10 days, 5 days in the preoperative period and 5 days in the postoperative period.
  Interventions: Other: The pre- and post- surgical breathing exercise group
- Control group (No Intervention): Routine practice group

INTERVENTIONS:
Other: The post-surgical breathing exercise group — Individuals in the Intervention-1 group were asked to perform 10 breathing exercises with IS every waking hour in addition to the routine practices of the clinic for 5 days in the postoperative period.
  Other Names: Intervention-1 group
  Arms: The post-surgical breathing exercise group
Other: The pre- and post- surgical breathing exercise group — Individuals in the Intervention-2 group were asked to perform 10 breathing exercises with IS every waking hour in addition to the routine practices of the clinic for a total of 10 days, 5 days in the preoperative period and 5 days in the postoperative period.
  Other Names: Intervention-2 group
  Arms: The pre- and post- surgical breathing exercise group

SUMMARY:
It was conducted as a single-center, prospective, randomized controlled experimental study. Data were collected with the Introductory Information Form, Numerical Rating Scale, Physiological Parameters Follow-up Form and General Comfort Scale.

DETAILED DESCRIPTION:
It was conducted as a single-center, prospective, randomized controlled experimental study. Data were collected with the Introductory Information Form, Numerical Rating Scale, Physiological Parameters Follow-up Form and General Comfort Scale.The study was conducted in three groups. Individuals in the intervention-1 group were asked to perform breathing exercises with IS in addition to the routine practices of the clinic for 5 days in the postoperative period. Individuals in the intervention-1 group were asked to perform breathing exercises with IS in addition to the routine practices of the clinic for a total of 10 days, 5 days in the preoperative period and 5 days in the postoperative period. Individuals in the control group were given only the routine practice of the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate in Turkish,
* undergoing cardiac surgery,
* no pain in the preoperative period (0 pain according to VA),
* have no problems with vision, hearing or speech,
* individuals who agreed to participate in the study were included.

Exclusion Criteria:

* Using psychiatric medication,
* Using immunosuppressive medication until 30 days before surgery,
* with neuromuscular disorders,
* having rheumatic disease,
* have had pulmonary surgery before,
* with cerebrovascular injury,
* diagnosed with cardiovascular instability or aneurysm,
* Diagnosed with COPD,
* individuals who do not volunteer to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-01-14 (Actual); Study Completion 2024-01-14 (Actual)

PRIMARY OUTCOMES:
Pain level | postop 1st and postop 5th day
  Evaluated with Numerical Rating Scale (NRS). NRS is a scale between 0 and 10.
Anxiety level | postop 1st and postop 5th day
  Evaluated with Numerical Rating Scale (NRS). NRS is a scale between 0 and 10.
Comfort level | postop 1st and postop 5th day
  It was evaluated with the General Comfort Scale. The scale is a four-point Likert type and contains a total of 48 items.
Partial oxygen pressure (PaO2) | postop 1st and postop 5th day
  It is evaluated with a sample taken from arterial blood.
Forced Vital Capacity (FVC) | postop 5th day
  It is measured with a device called spirometer.

CONTACTS AND LOCATIONS:
Overall Officials: SEVDA KORKUT, Principal Investigator — TC Erciyes University
Locations (1):
- Sevda Korkut, Talas, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No